CLINICAL TRIAL: NCT06636552
Title: An Investigator-Initiated, Phase II, Multicenter, Open-Label, Single-Arm, Prospective Clinical Trial to Evaluate the Efficacy and Safety of Alternating Bortezomib-Based Regimens in Combination With DaratUMumab Followed by Maintenance With Daratumumab in the Frontline Setting of Primary Plasma CEll LEukemIA: A Trial of the Greek Myeloma Study Group The " EUMELEIA " Study
Brief Title: An Investigator-Initiated, Phase II, Multicenter, Open-Label, Single-Arm, Prospective Clinical Trial to Evaluate the Efficacy and Safety of Alternating Bortezomib-Based Regimens in Combination With DaratUMumab Followed by Maintenance With Daratumumab in the Frontline Setting of Primary Plasma CEll L
Acronym: EUMELEIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Society of Hematology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54767414LEU2002
Record Dates: First submitted 2024-09-09; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Primary Plasma Cell Leukemia
Keywords: primary plasma cell leukemia
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: This is an investigator-initiated, prospective, multicenter, phase II, open-label, single-arm, non-randomized, single-stage clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Other): * A consolidation phase which includes two 21-day consolidation cycles of D-CVD
  * A maintenance phase which includes twenty-four 28-day cycles of daratumumab monotherapy (applicable for subjects who have achieved ≥PR at the end of consolidation phase [Cycle 8])
  Interventions: Drug: Daratumumab (Subcutaneously)

INTERVENTIONS:
Drug: Daratumumab (Subcutaneously) — D-PAD (21-Day Cycles 1, 3 and 5):
  1,800 mg (QW) SC on days 1, 8, and 15 (for Cycles 1 and 3) 1,800 mg (Q3W) SC on day 1 (for Cycle 5)
  D-CVD (21-Day Cycles 2, 4, 6, 7 and 8):
  1,800 mg (QW) SC on days 1, 8, and 15 (for Cycle 2) 1,800 mg (Q3W) SC on day 1 (for Cycles 4, 6, 7 and 8)
  Daratumumab monotherapy (28-Day Cycles 9 to 32):
  1,800 mg (Q4W) SC on day 1

SUMMARY:
The primary objective of this study is to evaluate the efficacy of the alternating D-PAD/D-CVD induction regimen followed by D-CVD consolidation regimen and maintenance with daratumumab monotherapy, in terms of PFS, in the first-line setting of pPCL.

DETAILED DESCRIPTION:
This is an investigator-initiated, prospective, multicenter, phase II, open-label, single-arm, non-randomized, single-stage clinical trial.

The study comprises the following phases:

A 28-day screening phase An induction phase which includes six 21-day induction treatment cycles of alternating D-PAD and D-CVD (starting with D-PAD) Note: Based on the post-induction treatment disease evaluation, transplant-eligible subjects who have achieved ≥SD and PBPC ≤2% will undergo ASCT whereas those with SD or PBPC 2% will discontinue study treatment. Accordingly, transplant-eligible subjects who have achieved ≥PR will receive 2 additional D-CVD cycles whereas those with <PR will discontinue study treatment.

ASCT (single or tandem) (applicable for transplant-eligible patients) A consolidation phase which includes two 21-day consolidation cycles of D-CVD A maintenance phase which includes twenty-four 28-day cycles of daratumumab monotherapy (applicable for subjects who have achieved ≥PR at the end of consolidation phase [Cycle 8]) An End of Treatment (EOT) visit: 30 days (±7 days) after the last dose of all components of the study treatment have been discontinued

A Post-Treatment Follow-Up (PTFU) phase which will begin once a subject permanently discontinues study treatment. In particular:

All subjects who complete or discontinue study treatment without disease progression (PD), will return to the site every 12 weeks (±2 weeks) for disease evaluation (or sooner at Investigator's discretion if there are concerns for progression/relapse) and other follow-up assessments until the earliest of confirmed PD, start of subsequent therapy for PCL, death, or the end of study (EOS) definition is met.

After confirmed PD or the start of a new anticancer treatment for PCL, subjects will return to the site or be contacted by telephone every 16 weeks (±2 weeks) for collection of follow-up information (i.e., other malignancies, next-line therapy, and survival, as applicable) until death, withdrawal of consent for study participation, or the EOS definition is met, whichever occurs first.

ELIGIBILITY:
Inclusion

1. Age between 18 and 80 years (inclusive) at the time of signing the informed consent.
2. Patients newly diagnosed with documented pPCL as defined by the current IMWG criteria for PCL and MM:

   * Documented presence of ≥5% PBPCs and/or absolute number ≥0.5 × 103/μL, assessed either morphologically in the peripheral blood (PB) smear or by flow cytometry, and confirmation of plasma cell clonality by flow cytometry
   * Clonal BMPCs ≥10% or biopsy-proven bony or extramedullary plasmacytoma
   * At least one of the following myeloma defining events:
   * Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically (one or more of the following):
   * Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than the upper limit of normal (ULN) or >2.75 mmol/L (>11 mg/dL)
   * Renal insufficiency: Creatinine clearance (CrCl) <40 mL/min (measured or estimated by validated equations) or serum creatinine >177 μmol/L (>2 mg/dL)
   * Anemia: hemoglobin value of >20 g/L below the lower limit of normal (LLN), or a hemoglobin value <100 g/L
   * Bone lesions: One or more osteolytic lesions on skeletal radiography, computed tomography (CT), or positron emission tomography (PET)-CT.
   * Any one or more of the following biomarkers of malignancy:
   * Clonal bone marrow plasma cell percentage ≥60%
   * Involved:Uninvolved serum free light chain (sFLC) ratio ≥100 >1 focal lesions on MRI studies (each focal lesion must be 5 mm or more in size).
3. Measurable disease by protein electrophoresis as defined by any of the following:

   * Serum M-protein level:
   * For IgG MM: ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours
   * For IgA, IgE and IgM MM: ≥0.5 g/dL or urine M-protein level ≥200 mg/24 hours
   * For IgD MM: ≥0.05 g/dL or urine M-protein level ≥200 mg/24 hours
   * Light chain MM without measurable disease in the serum or the urine: sFLC ≥10 mg/dL (involved light chain) and abnormal sFLC κ/λ ratio.
4. Patients for whom high-dose therapy, with or without stem cell transplantation, is part of the intended treatment plan.
5. Patient not currently or previously treated with any systemic therapy or stem cell transplant for any plasma cell dyscrasia, apart from a short course of corticosteroid therapy (equivalent of dexamethasone 40 mg/day for up to 4 days).
6. Adequate bone marrow function as determined by the following:

   * Hemoglobin ≥7.0 g/dL [≥4.34 mmol/L; prior red blood cell transfusion or recombinant human erythropoietin use is permitted]
   * Absolute neutrophil count ≥1.0 x 109/L [granulocyte-colony stimulating factor use is permitted]
   * Platelet count ≥50 x 109/L if disease involvement in bone marrow is >50%; otherwise ≥75% x 109/L.
7. Adequate liver function as determined by the following:

   * Serum Aspartate Transaminase ≤2.5 x ULN
   * Serum Alanine Aminotransferase ≤2.5 x ULN
   * Total bilirubin ≤1.5 x ULN (for subjects with congenital bilirubinemia, such as Gilbert syndrome, direct bilirubin ≤1.5 x ULN is required).
8. Adequate renal function as determined by estimated CrCl ≥20 mL/min.
9. Eastern Cooperative Oncology Group (ECOG) Performance status 0-3.
10. If females of childbearing potential (FCBP), the following apply:

    * Willingness to use an acceptable form of birth control during the clinical trial. FCBPs must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously during the treatment period, and for 3 months after the last dose of any component of the treatment regimen.
    * They must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 3 months after receiving the last dose of any component of the study treatment.
    * They must have 2 negative serum or urine pregnancy tests; one at Screening and in particular within 10-14 days prior to C1D1, and the second within 24 hours prior to C1D1.
11. If male subjects of reproductive potential who are sexually active with FCBPs the following apply.

    * Must always use a latex or synthetic condom during the study and for 3 months after discontinuing study treatment (even if they have undergone a successful vasectomy).
    * They must not donate sperm during the study or for 3 months after the last dose of study treatment.
12. Patients who are able to comprehend and willing to follow the requirements of the study.
13. Patients (or patients' legally acceptable representative as applicable) who are able to understand and willing to provide voluntary written informed consent before any clinical trial-related procedure is performed.

Exclusion

1. Patients with secondary PCL.
2. Prior or concurrent invasive malignancy (other than PCL) within 5 years of date of study treatment initiation except for the following:

   * Malignancy treated with curative intent and with no known active disease present for ≥3 years before study treatment initiation.
   * Adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix or breast, incidental histologic finding of prostate cancer (T1a or T1b) or other non-invasive lesion that, as per Investigator's judgement, is considered cured with minimal risk of recurrence over the next 3 years.
3. Radiation therapy within 14 days before study treatment initiation.
4. Plasmapheresis within 28 days before study treatment initiation.
5. Exhibiting clinical signs of meningeal or central nervous system involvement by PCL.
6. Patients with peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.
7. Concurrent systemic amyloidosis, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and/or skin changes), active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease, and any other medical condition/disease that is likely to interfere with the study procedures or results, or that in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
8. Known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second [FEV1] <50% of predicted normal.
9. Known moderate or severe persistent asthma within the past 2 years, or the patient currently has uncontrolled asthma of any classification.
10. Any of the following:

    * Known seropositivity for human immunodeficiency virus
    * Seropositivity for hepatitis B virus defined by a positive test for hepatitis B surface antigen.
    * Known seropositivity for hepatitis C virus defined by anti-HCV antibody positive or HCV-RNA quantitation positive.
11. Clinically significant cardiac disease including:

    * Myocardial infarction within 6 months before study treatment initiation
    * Unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV)
    * Pericardial disease
    * Cardiac amyloidosis
    * Uncontrolled cardiac arrhythmia (NCI CTCAE v5 Grade 2 or higher) or clinically significant electrocardiogram (ECG) abnormalities
    * Screening 12-lead ECG showing a baseline QT interval >470 msec (except for subjects with pacemaker)
    * Screening transthoracic echocardiogram showing left ventricular ejection fraction (LVEF) <40% (screening TTE is required only for subjects aged ≥ 65 years).
12. Receipt of a strong CYP3A4 inducer within 5 half-lives prior to study treatment initiation.
13. Known allergies, hypersensitivity, or intolerance to boron or mannitol, corticosteroids, monoclonal antibodies or human proteins, or their excipients, or known sensitivity to mammalian-derived products.
14. Gastrointestinal disease that may significantly affect the absorption of oral drugs as per Investigator's discretion.
15. Vaccination with live attenuated vaccines within 4 weeks of study treatment initiation.
16. Major surgery within 2 weeks before study treatment initiation or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to start the study treatment.
17. Concurrent use of other anti-cancer agents/treatments.
18. Subject is known or suspected of not being able to comply with the study protocol (e.g., because of alcoholism, drug dependency, or psychological disorder). Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
19. Females who are pregnant, breast feeding, or planning to become pregnant while enrolled in this study or within 3 months following the last dose of any component of the study treatment.
20. Males who plan to father a child while enrolled in this study or within 3 months following the last dose of any component of the study treatment.
21. Patients who currently receive treatment with any investigational drug/vaccine/device/intervention or who have received any investigational product within 30 days or 5 half-lives of the investigational agent (whichever is longer) before the screening.
22. Contraindications to the use of any components of the study treatment (daratumumab, bortezomib, dexamethasone, cyclophosphamide, doxorubicin) per local prescribing information.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2029-01-05 (Estimated); Study Completion 2029-01-05 (Estimated)

PRIMARY OUTCOMES:
Εfficacy of the alternating D-PAD/D-CVD induction regimen followed by D-CVD consolidation regimen and maintenance with daratumumab monotherapy, in terms of PFS, in the first-line setting of pPCL. | Approximately 28 months (including induction/consolidation/maintenance phase and excluding transplantation) [168 days induction/consolidation plus 672 days maintenance].
  Duration from the date of induction treatment initiation to the date of first documented evidence of progressive disease (PD) (assessed by the IMWG criteria) or death, whichever occurs earlier.

CONTACTS AND LOCATIONS:
Locations (7):
- Greece (7):
  - 1st Propaedeutic Department, "Laiko" General Hospital of Athens, Athens, Attica
  - Hematology Clinic, General Hospital of Athens "Evanggelismos", Athens, Attica
  - Hematology Department "Alexandra" General Hospital of Athens, Athens, Attica
  - Hematology Department, University General Hospital of Alexandroupolis, Alexandroupoli, Evros
  - Hematology Department, Regional General Hospital for Cancer Treatment "Metaxa" of Piraeus, Piraeus
  - Hematology Department, General Hospital of Thessaloniki "Papanikolaou", Thessaloniki
  - Hematology Department, Theageneion Cancer Hospital, Thessaloniki